CLINICAL TRIAL: NCT03103269
Title: Challenge! in Baltimore City Middle Schools
Brief Title: Challenge! Adolescent Obesity Prevention
Acronym: Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Johns Hopkins Bloomberg School of Public Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00040540; R01HD054727 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2017-04-06 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Prevention; Diet; Physical activity; Depression; Anxiety; Stages of change; Barriers; Perceptions; Environment; Eating Disorder; Self efficacy
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Depression; Anxiety Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Challenge! Small Group Intervention only (Experimental): This group receives the Challenge! Small Group intervention consisting of curriculum related to health behavior goal setting, healthy eating, and staying active, works out with their Health Educators, and receives a year-long membership to the YMCA.
  This group is in schools that were randomly assigned to NOT receive the Environmental Intervention.
  Interventions: Behavioral: Challenge! Small Group Intervention
- Challenge! Small Group and Environmental Intervention (Experimental): This group consists of participants who receive the Challenge! Small Group Intervention AND attend a school that is randomly assigned to receive an environmental intervention.
  This group receives the Challenge! Small Group intervention consisting of curriculum related to health behavior goal setting, healthy eating, and staying active, works out with their Health Educators, and receives a year-long membership to the YMCA.
  The environmental intervention involves the formation of a Health and Activity Committee composed of community members, teachers, parents, school staff, and 8th grade girls from the school. Together, this group comes up with ways to make their school environment healthier.
  Interventions: Behavioral: Challenge! Small Group Intervention; Other: Challenge! Environmental Intervention
- Environmental Intervention Only (Experimental): This group consists of participants who do not receive the Challenge! Small Group Intervention but attend a school that is randomly assigned to receive an environmental intervention.
  This group does not receive the Challenge! Small Group Intervention.
  The environmental intervention involves the formation of a Health and Activity Committee composed of community members, teachers, parents, school staff, and 8th grade girls from the school. Together, this group comes up with ways to make their school environment healthier.
  Interventions: Other: Challenge! Environmental Intervention
- Control Group (No Intervention): This group does not receive the Challenge! Small Group intervention and is in a school that is randomly assigned to NOT have the Environmental Intervention.

INTERVENTIONS:
Behavioral: Challenge! Small Group Intervention — The Challenge! Small Group intervention consists of curriculum related to health behavior goal setting, healthy eating, and staying active, working out with Health Educators, and receiving a year-long membership to the YMCA.
  Arms: Challenge! Small Group Intervention only; Challenge! Small Group and Environmental Intervention
Other: Challenge! Environmental Intervention — The environmental intervention involves the formation of a Health and Activity Committee composed of community members, teachers, parents, school staff, and 8th grade girls from the school. Together, this group comes up with ways to make their school environment healthier.
  Arms: Challenge! Small Group and Environmental Intervention; Environmental Intervention Only

SUMMARY:
The prevalence of overweight among adolescents (BMI-for-age %tile over the 95th percentile) has more than tripled over the past 3 decades in the US. Overweight and physical inactivity disproportionately affect low- income, female, African American adolescents.

A prior health-promotion/ obesity-prevention program for adolescents developed and tested by our group (Challenge!) showed that adolescents who received the intervention were less likely to become overweight or obese over 2 years when compared to the control group. This intervention was administered one-on-one to adolescents in their homes or community by a college-aged mentor.

Schools are an ideal setting for interventions because the effect can be far-reaching and sustainable. School-based obesity-prevention interventions have thus far shown modest results.

The purpose of this study is to evaluate the impact of a multilevel intervention that includes both the Challenge program administered in a small group format after school using mentors and teachers and a school-wide environmental change on adolescent females' body composition, diet, and physical activity. The intervention is targeted to 6th and 7th grade female students. The small group intervention is conducted over 12 weeks and includes goal setting focusing on healthy diet and physical activity, along with membership and weekly trips to the YMCA. The environmental intervention includes a Health and Activity Committee (HAC), comprised of 8th grade female students (popular opinion leaders), school personnel, parents, and community members. The HAC develops school-wide health promotion messages and activities. Parents of participating 6th and 7th grade girls provide information on family variables. The hypotheses are that females who receive the small group or environmental intervention are at less risk of weight gain (overweight) than females in the control small group condition, that females in environmental schools are at less risk of weight gain (overweight) than females in the control environmental condition, and that females who receive both the small group and environmental intervention are at the lower risk of weight gain (overweight) than females who receive only the environmental or small group intervention or neither intervention.

ELIGIBILITY:
Inclusion Criteria:

For small group intervention:

* Female Adolescent
* Grades 6 or 7
* No health problems that would interfere with participation in physical education classes

For environmental intervention Health and Activity Committee:

Must be one of the following:

* 8th grade female student
* Parent or legal guardian of any student in the school
* School personnel
* Adult Community member (Self-identifies as member of specified community surrounding school)

Exclusion Criteria:

For small group intervention:

* Male
* Outside of the grade range 6-7 at recruitment
* Participant will be excluded if they answer no to question 1 on the screening questionnaire (unable to read and understand questions written in English)
* Participant will be excluded if they answer yes to questions 2 or 3 on screening form (fails health screening due to medical condition preventing them from engaging in physical activity)

For environmental intervention Health and Activity Committee:

* Inability to speak or read English
* Inability to attend meetings

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change of Body Mass Index Percentile for Age and Sex for adolescent females | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up

SECONDARY OUTCOMES:
Change of Dietary Quality for adolescent females | Baseline to 6 month (Post Intervention) Follow-up or 1 year (Delayed Intervention) Follow-up
  Dietary quality will be assessed via the use of a Food Frequency Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, PhD, Principal Investigator — University of Maryland School of Medicine, Department of Pediatrics, Growth & Nutrition Division
Locations (1):
- Baltimore City Public Schools, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Trude ACB, Armstrong B, Kramer Fiala Machado A, Wickwire EM, Covington LB, Wang Y, Hager E, Black MM. Waking up to sleep's role in obesity and blood pressure among Black adolescent girls in low-income, US urban communities: A longitudinal analysis. Sleep Health. 2022 Apr;8(2):200-207. doi: 10.1016/j.sleh.2021.12.001. Epub 2022 Feb 11. PMID 35153168